CLINICAL TRIAL: NCT01443767
Title: Pilot Study to Examine the Correlation of 'Estimated Continuous Cardias Output' (esCCO) With Pulse Contour Analysis of the Arterial Waveform (Picco) in Partial Liver Resection
Brief Title: Correlation of Estimated Continuous Cardias Output (esCCO) and Picco in Partial Liver Resection
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: Nihon Kohden Europe (Unknown)
Responsible Party: Principal Investigator, Christoph Schramm, M.D., Principal Investigator, Heidelberg University
Other Study IDs: S188/2011
Record Dates: First submitted 2011-09-26; First posted 2011-09-30 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Continuous Cardiac Output
Keywords: Cardiac Output; esCCO; Pulse Wave Transit Time; PiCCO; Pulse Contour Analysis; Non-invasive Monitoring; Partial Liver Resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Partial liver resection: Adult patients scheduled for elective partial liver resection

SUMMARY:
The purpose of this study is to determine the measuring accuracy of the truly non-invasive method estimated continuous cardiac output (esCCO) against the reference method pulse contour analysis of the arterial waveform (Picco) in partial liver resection. esCCO is calculated using the pulse wave transit time, which is defined as the time between the R-wave of the ECG and a 30% increase of the differentiated pulseoximetry waveform.

DETAILED DESCRIPTION:
The objective is to compare two methods of cardiac output measurement: the new non-invasive method called esCCO™ (by Nihon Kohden, Tokyo, Japan) and the established more invasive method PiCCO™ (by PULSION Medical Systems, Munich, Germany). esCCO™ is a completely non-invasive method that could provide a cardiac output measurement in a large range of patients because of an extremely low risk benefit balance. Thus the valuable information of cardiac output in combination with standard patient monitoring could be integrated in the assessment and clinical handling of a patients circulatory system.

In previous Japanese studies, esCCO™ was tested against the pulmonary artery catheter in patients undergoing heart surgery. Because of promising results in those studies, the validity of the method is now tested in patients scheduled for partial liver resection as a major visceral surgery intervention. Partial liver resection is a medium to high risk surgical intervention because of the extended blood supply of the organ. High and sudden blood loss can easily occur during the operation. Measurement period starts at the beginning of anesthesiologic induction and is continued until the extubation at the end of the intervention.

The algorithm for esCCO™ -measurement is integrated in an approved patient monitor that replaces the standard patient monitor during the measurement-period. The PiCCO™-device is added on the same rack and a cable connects the PiCCO™-device to the patient monitor. To assure maximum quality of the reference method, a thermodilution for PiCCO™-calibration is accomplished every 30 minutes.

In the study protocol, events like esCCO™ - and PiCCO™-calibration time, catheter positioning time, changes of the patient's position, ventilation settings, volume in- and output and drug administration, patients's data and diagnoses are logged. Vital parameters from the patient monitor including the PiCCO™-cardiac output values are recorded every second in real time on a study laptop mounted on the same rack as the patient monitor and the PiCCO™ device but separated electrically from the other devices.

A total of 30 patients shall be investigated in the study during a planned study time of approximately 6 months. The ethics committee of the University of Heidelberg gave their consent to the study (S-188/2011). The investigators will approximately receive 1080 data pairs when averaging the values every 5 minutes with a mean duration of the surgical procedure of 3 hours.

For statistical analysis, a Bland-Altman-test for multiple values in one patient, a t-test for depending values, correlation graphics and a regression equation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* patient scheduled for partial liver resection
* sinus rhythm

Exclusion Criteria:

* no written consent
* continuous severe cardiac arrhythmias
* cardiac pacemaker
* intraaortal balloon pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients scheduled for partial liver resection
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Correlation of esCCO and Picco in Partial Liver Resection | Intraoperative (Measurement from induction of anaesthesia to extubation)

CONTACTS AND LOCATIONS:
Overall Officials: Konstanze Plaschke, Professor, Study Chair — Heidelberg University; Christoph Schramm, M.D., Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany